CLINICAL TRIAL: NCT00308243
Title: Inhaled Sodium Pyruvate for the Treatment of Cystic Fibrosis. A Phase I, Double Blind, Placebo Controlled, Safety Study. Stage 1)
Brief Title: Inhaled Sodium Pyruvate for the Treatment of Cystic Fibrosis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emphycorp (Industry)
Collaborators: Cellular Sciences, inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSI-N115-I-010-01; Orphan Drug 02-1656
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Sodium Pyruvate; Reactive Oxygen Species; Inflammation of Lung
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sodium Chloride

INTERVENTIONS:
Drug: Sodium Pyruvate in 0.9% Sodium Chloride Solution

SUMMARY:
It is hypothesized that the inhalation of sodium pyruvate will reduce lung damage in patients with Cystic Fibrosis (CF) by its ability to reduce levels of toxic reactive oxygen and nitrogen compounds associated with the chronic inflammatory component of the disease. The primary objective of the study is to assess the safety of inhaled sodium pyruvate in 0.9% sodium chloride (saline) solution in people with CF. Further, to determine whether inhaled sodium pyruvate will improve lung function, as determined by spirometry, or reduced inflammatory markers in induced sputum of people with CF.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common, lethal inherited disease of Caucasians. Approximately 30,000 people in the United States and 70,000 worldwide have a diagnosis of CF. It is caused by mutations in the cystic fibrosis transmembrane regulator (CFTR) gene. The clinical manifestations characteristic of CF include progressive bronchiectatic lung disease with thick mucus production and colonization by Pseudomonas aeruginosa. The CFTR gene mutation results in altered cell transport properties, which affect both chloride and glutathione secretion. Chronic inflammation, associated with activated neutrophils and macrophages, is a common feature of CF. Highly reactive toxic oxygen (superoxide anion, free hydroxyl radical, hydrogen peroxide) and nitrogen species (nitric oxide, peroxynitrites) are abundant in the chronic inflammatory response in CF and appear to play a prominent role in the pathogenesis of this disease. These reactive oxygen and nitrogen species have been shown to be directly toxic to various mammalian tissues, including lung, via DNA damage and cell membrane lipid peroxidation. In addition, elevated levels of hydrogen peroxide and nitric oxide have been demonstrated in sputum and bronchoalveolar lavage fluid of patients with CF, asthma, and chronic obstructive pulmonary disease. Clearly reactive oxygen and nitrogen species are implicated in the pathogenesis of a variety of lung diseases including CF.

Sodium pyruvate is an antagonist of both reactive oxygen and nitrogen species. It also has the potential to increase intracellular levels of thiol compounds, major sources of intracellular anti-oxidants. Sodium pyruvate has been shown to act as an anti-inflammatory agent that can reduce the number of infiltrating neutrophils and levels of oxygen radicals at wound sites, thereby limiting the production of pro-inflammatory mediators. Thus, it is hypothesized that the inhalation of sodium pyruvate will reduce lung damage in patients with CF by its ability to reduce levels of toxic reactive oxygen and nitrogen species associated with the chronic inflammatory component of the disease.

The trial is a Phase I Safety Study that will be conducted in three Stages. The study is designed to assess the safety of administering sodium pyruvate inhalation therapy to CF subjects once a day for one day, then twice a day for one day, and finally, twice a day for four weeks. All testing, including the screening visit and Stage 1, and Stages 2 and 3, will be conducted at the University of Minnesota (UMN) General Clinical Research Center GCRC).

Stage 1 - Single dose inhalation - 24 hours (n=15) Participants with CF will receive a single dose of sodium pyruvate (5 ml in physiological saline) via a Pari-Jet hand-held nebulizer (Pari LC Plus® nebulizer system) , and will be followed at UMN GRC for four hours with a follow up telephone interview at 24 hours. Three concentrations (0.5 mM, 1.5 mM, and 5.0 mM) of sodium pyruvate solution will be studied. Five subjects will receive the lowest concentration of sodium pyruvate solution; then another five subjects will receive the middle dose of sodium pyruvate solution; and finally a third group of five subjects will receive the highest dose of sodium pyruvate solution.

Patients enrolled in Stage 1 will have one 6-hour visit at UMN GCRC. Following administration of a single 5-mL dose of either 0.5 mM, 1.5 mM, or 5.0 mM sodium pyruvate in 0.9% saline solution, the following tests will be performed:

Post Inhalation of Study Drug

Spirometry:

* Post inhalation 0.5 Hr
* Post inhalation 1 Hr
* Post inhalation 2 Hr
* Post inhalation 4 Hr

Sputum Induction:

* Post inhalation 1 Hr

SaO2:

* Post inhalation 0.5 Hr
* Post inhalation 1 Hr
* Post inhalation 2 Hr
* Post inhalation 4 Hr

End of Visit.

Blood and Urine Analysis

* Post inhalation 4 Hr

Electrocardiogram

* Post inhalation 4 Hr

Vital Signs

* Post inhalation 4 Hr

The parameters for safety monitoring will include spirometry, vital signs, ECG, SaO2, and routine blood and urine analysis, which will be conducted pre- and post- inhalation of sodium pyruvate. Follow up telephone interviews will also be conducted for each stage.

With regard to efficacy, spirometry, and induced sputum samples will be monitored pre- and post- inhalation of sodium pyruvate. Induced sputum samples will be evaluated for cellular content (total WBC and differential) and the fluid content assessed for total protein, total DNA, elastase, glutathione (GSH and GSSG), H2O2 and inflammatory cytokines (IL-1, IL-6, and IL-8, TNF-alpha).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CF using Cystic Fibrosis Foundation criteria.
* FEV1 >40% predicted
* Colonization with Pseudomonas aeruginosa - (>= 2 positive cultures over past 12 months)
* >18 years of age
* Stable respiratory status without dyspnea
* Non-smoker
* Able to perform sputum induction

Exclusion Criteria:

* Severe CF with an FEV1 of <40% predicted
* Lung disease not CF related
* Positive culture for Burkholderia cepacia
* Active allergic bronchopulmonary aspergillosis
* Clinically significant cardiac disease
* Pregnancy
* Females of child bearing age not using contraception
* Females lactating
* <18 years of age
* Systemic steroid treatment within 1 month
* Hospitalization within 3 months due to airway disease
* Immunotherapy
* Changes in respiratory medication use within 1 month
* New medications within 1 month
* Participation in research study within 1 month
* History of significant (>60 cc) hemoptysis within 1 year
* Poorly controlled insulin dependent diabetes mellitus
* Acute respiratory illness within 1 month
* Use of tobacco products or recreational drugs
* History of adverse reaction to sputum induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable is the assessment of safety of inhaled sodium pyruvate in subjects with CF.

SECONDARY OUTCOMES:
The secondary outcome variable is the determination of improvement in lungs of CF subjects as determined by measurement of FEV1 and/or as determined by measurement of reduced inflammatory markers in induced sputum.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Billings, MD, Study Director — University of Minnesota; Pulmonary, Allergy & Critical Care Medicine
Locations (1):
- University of Minnesota Medical School, The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota, United States

REFERENCES:
- See also: Click here for more information about this study: Inhaled Sodium Pyruvate for the Treatment of Cystic Fibrosis. A Phase I, Double Blind, Placebo Controlled, Safety Study. (Stage 1) — http://www.emphycorp.com/